CLINICAL TRIAL: NCT00669643
Title: Independent Study to Establish the Efficacy of the Six Doses Uniform MDT Regimen (U-MDT) for Leprosy Patients
Brief Title: Uniform Multidrug Therapy Regimen for Leprosy Patients
Acronym: U-MDT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Brasilia (Other)
Collaborators: Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government); Ministry of Science and Technology, Brazil (Other); Ministry of Health, Brazil (Other Government); Fundação Alfredo da Matta, Manaus, Brazil (Unknown); Instituto de Dermatologia Dona Libania, Fortaleza, Brazil (Unknown)
Responsible Party: Principal Investigator, Gerson Oliveira Penna, Dr., University of Brasilia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNPq / DECIT 403293/2005-7
Record Dates: First submitted 2008-04-24; First posted 2008-04-30 (Estimated); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Leprosy
Keywords: Leprosy; Communicable Diseases; Skin Diseases; Multidrug Therapy; MDT; Uniform Multidrug Therapy; U-MDT
MeSH Terms: conditions — Leprosy; Communicable Diseases; Skin Diseases | interventions — Rifampin; Dapsone; Clofazimine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- R-MDT PB (Active Comparator): R-MDT PB group: standard/regular treatment recommended by WHO - All patients presenting fewer than 6 skin lesions will receive the standard treatment regimen for paucibacillary patients as the intervention; Intervention - PB 6 doses of rifampicin and dapsone
  Interventions: Drug: PB 6 doses - Rifampicin and Dapsone
- U-MDT PB (Experimental): U-MDT PB group: a unified treatment for all patients - All patients presenting fewer than 6 lesions (WHO PB) will receive 6 doses of rifampicin, clofazimine and dapsone as the intervention; Intervention - PB 6 doses of rifampicin, clofazimine and dapsone
  Interventions: Drug: PB 6 doses - Rifampicin, Clofazimine and Dapsone
- R-MDT MB (Experimental): R-MDT MB group: standard/regular treatment recommended by WHO - All patients presenting 6 skin or more lesions will receive the standard treatment regimen for multibacillary patients as the intervention; Intervention - MB 12 doses of rifampicin, clofazimine and dapsone
  Interventions: Drug: MB 12 doses - Rifampicin, Clofazimine and Dapsone
- U-MDT MB (Experimental): U-MDT MB group: a unified treatment for all patients - All patients presenting 6 lesions or more (WHO MB) will receive 6 doses of rifampicin, clofazimine and dapsone as the intervention; Intervention - MB 6 doses of rifampicin, clofazimine and dapsone
  Interventions: Drug: MB 6 doses - Rifampicin, Clofazimine and Dapsone

INTERVENTIONS:
Drug: PB 6 doses - Rifampicin and Dapsone — Adult: 6 doses;
  1 monthly supervised dose: 600 mg Rifampicin + 100 mg Dapsone; 27 days: p/day - 100 mg Dapsone;
  Children: 6 doses;
  1 monthly supervised dose: 450 mg Rifampicin + 50 mg Dapsone; 27 days: p/day - 50 mg Dapsone
  Other Names: PB 6 doses of 2 drugs
  Arms: R-MDT PB
Drug: PB 6 doses - Rifampicin, Clofazimine and Dapsone — Adult: 6 doses;
  1 monthly supervised dose: 600 mg Rifampicin + 300 mg Clofazimine + 100 mg Dapsone; 27 days: p/day - 100 mg Dapsone + 50 mg Clofazimine;
  Children: 6 doses;
  1 monthly supervised dose: Rifampicin 450 mg + 150 mg Clofazimine + 50 mg Dapsone; 27 days: p/day - 50 mg Dapsone + 25 mg Clofazimine
  Other Names: PB 6 doses of 3 drugs
  Arms: U-MDT PB
Drug: MB 12 doses - Rifampicin, Clofazimine and Dapsone — Adult: 12 doses;
  1 monthly supervised dose: 600 mg Rifampicin + 300 mg Clofazimine + 100 mg Dapsone; 27 days: p/day - 100 mg Dapsone + 50 mg Clofazimine;
  Children: 12 doses;
  1 monthly supervised dose: Rifampicin 450 mg + 150 mg Clofazimine + 50 mg Dapsone; 27 days: p/day - 50 mg Dapsone + 25 mg Clofazimine
  Other Names: MB 12 doses of 3 drugs
  Arms: R-MDT MB
Drug: MB 6 doses - Rifampicin, Clofazimine and Dapsone — Adult: 6 doses
  1 monthly supervised dose: 600 mg Rifampicin + 300 mg Clofazimine + 100 mg Dapsone; 27 days: p/day - 100 mg Dapsone + 50 mg Clofazimine
  Children: 6 doses
  1 monthly supervised dose: Rifampicin 450 mg + 150 mg Clofazimine + 50 mg Dapsone; 27 days: p/day - 50 mg Dapsone + 25 mg Clofazimine
  Other Names: MB 6 doses of 3 drugs
  Arms: U-MDT MB

SUMMARY:
The purpose of this randomized trial is to verify if leprosy patients, despite of their classification, can be treated with the same regimen without compromising patient cure and acceptability of the treatment. At present, patients classified as multibacillary leprosy are treated for 12 months with three drugs, and patients classified as paucibacillary leprosy are treated for 6 months with two drugs. The study is going to test a unified regimen for paucibacillary and multibacillary patients by treating leprosy patients with three drugs for 6 doses.

DETAILED DESCRIPTION:
In the past both the treatment of new leprosy patients and the classification criteria for treatment purposes have gone through major changes. At the moment, newly diagnosed leprosy patients are classified into PB and MB based on the number of lesions only. More than 5 lesions leads to a classification as MB patient and treatment for 12 months with MDT composed of three drugs, i.e. rifampicin, dapsone and clofazimine. One to 5 lesions leads to a classification as PB patient and treatment for 6 months with MDT composed of two drugs, i.e. rifampicin and dapsone.

Despite all the favorable data from the point of view of practical application, this therapeutic regimen still presents some constraints, including the lengthy course of treatment. Especially in those situations where leprosy control is integrated into the general health services classification is a problem for the general health worker that has only received one or two days of training in leprosy.

A uniform regimen for leprosy would simplify treatment in the field. Results from control programs and research projects have demonstrated that relapse rates after MDT are extremely low, approximately 0.2% annually among MB cases on the 24-dose regimen. The low relapse rates indicate that there was room to shorten the course of MDT to less than 24 monthly-supervised doses of rifampicin plus self-administered doses of dapsone and clofazimine. Although some papers have suggested that relapse rates after MDT may be significantly higher in MB patients with an initial bacterial index equals or bigger than 3, the present diagnostic universe of leprosy includes few such patients, and the total number of relapses caused by them would account for a minimal percentage of cases in a control program. Since 1998, a 12-month treatment course for MB leprosy is advised by WHO. The main problem when evaluating any new treatment regimen for leprosy, is that there are no good and reliable data available for the current treatment regimen: relapse rates have never been systematically determined and the same holds true for reaction and nerve function impairment rates, the major cause of the nerve damage that leads to handicaps and deformities in leprosy patients.

Currently, WHO is exploring possibilities to introduce a short uniform treatment regimen for all types of leprosy patients called Uniform Multidrug Therapy (U-MDT), as a replacement for the present regular multidrug therapy (R-MDT). This U-MDT would consist of treatment of all patients for 6 months with a regimen consisting of three drugs: rifampicin, dapsone and clofazimine. The efficacy of this U-MDT is currently being studied in an open non-controlled treatment trial. Classification of patients is only done on clinical criteria: no skin smears or other lab tests are included. The diagnosis of relapse will rely on clinical diagnosis only. It will therefore not be possible to identify high-risk groups for relapse, such as highly skin smear positive patients.

The objective of our study is to evaluate both the R-MDT and the U-MDT regimens in a randomised trial in order to:

1. determine the efficacy of the current R-MDT regimen with regard to relapse rates and acceptability to the patient.
2. determine the efficacy of the U-MDT regimen with regard to relapse rate and acceptability to the patient.

ELIGIBILITY:
Inclusion Criteria:

* All newly diagnosed leprosy cases with characteristic skin lesions, with or without systemic symptoms or confirmed by histopathological study previously untreated PB and MB leprosy patients.
* Never treated or patient treated more than five years ago

Exclusion Criteria:

Safety concerns:

* History of intolerance to one of the medications

Lack of suitability for the trial:

* Absence of leprosy skin lesions
* Pure neural leprosy (PNL)
* Patient previously (defaulters and relapse) treated for leprosy less than 5 years ago
* Association with other serious diseases such as HIV/AIDS, Tuberculosis, Malaria, American Cutaneous leishmaniasis, Visceral Leishmaniasis, Lymphoma, Leukaemia, Immunosuppression, etc.

Administrative reasons

* Patients who are not permanent residents of the area or who are unable to come to the clinic every month during their treatment and in the first half year (the intensive follow-up period) after their treatment.
* Patients who do not give informed consent or are not capable to give informed consent due to mental impairment.
* Patients with overt signs of AIDS because it is unlikely that we can follow them up for the whole study period. As we will not be testing patients for HIV positivity, HIV-infected leprosy patients can be included in the study.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 859 (Actual)
Dates: Start 2007-02; Primary Completion 2012-09 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Relapse | 5 years

SECONDARY OUTCOMES:
Type I Reaction - Reversal Reactions | 6 years
Type II Reaction - Erythema nodosum leprosum | 6 years
Neurological damage | 6 years
Neuritis | 6 years

CONTACTS AND LOCATIONS:
Overall Officials: Gerson O Penna, MD, PhD, Principal Investigator — University of Brasilia; Samira Buhrer, PhD, Study Director — Federal University of Goiás
Locations (2):
- Brazil (2):
  - Centro de Referência Nacional Alfredo da Matta - FUAM, Manaus, Amazonas
  - Centro de Referência Nacional Dona Libânia - CDERM, Fortaleza, Ceará

IPD SHARING:
Plan to Share IPD: No
Data sharing was not previously requested to the Ethical Committee. Therefore, if there will be a request for it, new ethical approval must be obtained.

REFERENCES:
- [Background] Becx-Bleumink M. Relapses among leprosy patients treated with multidrug therapy: experience in the leprosy control program of the All Africa Leprosy and Rehabilitation Training Center (ALERT) in Ethiopia; practical difficulties with diagnosing relapses; operational procedures and criteria for diagnosing relapses. Int J Lepr Other Mycobact Dis. 1992 Sep;60(3):421-35. PMID 1474281
- [Background] Britton WJ, Lockwood DN. Leprosy. Lancet. 2004 Apr 10;363(9416):1209-19. doi: 10.1016/S0140-6736(04)15952-7. PMID 15081655
- [Background] Buhrer-Sekula S, Smits HL, Gussenhoven GC, van Leeuwen J, Amador S, Fujiwara T, Klatser PR, Oskam L. Simple and fast lateral flow test for classification of leprosy patients and identification of contacts with high risk of developing leprosy. J Clin Microbiol. 2003 May;41(5):1991-5. doi: 10.1128/JCM.41.5.1991-1995.2003. PMID 12734239
- [Background] Dasananjali K, Schreuder PA, Pirayavaraporn C. A study on the effectiveness and safety of the WHO/MDT regimen in the northeast of Thailand; a prospective study, 1984-1996. Int J Lepr Other Mycobact Dis. 1997 Mar;65(1):28-36. PMID 9207751
- [Background] Jamet P, Ji B. Relapse after long-term follow up of multibacillary patients treated by WHO multidrug regimen. Marchoux Chemotherapy Study Group. Int J Lepr Other Mycobact Dis. 1995 Jun;63(2):195-201. PMID 7602214
- [Background] Jesudasan K, Vijayakumaran P, Manimozhi N, Jeyarajan T, Rao PS. Absence of relapse within 4 years among 34 multibacillary patients with high BIs treated for 2 years with MDT. Int J Lepr Other Mycobact Dis. 1996 Jun;64(2):133-5. PMID 8690971
- [Background] Li HY, Hu LF, Wu PW, Luo JS, Liu XM. Fixed-duration multidrug therapy in multibacillary leprosy. Int J Lepr Other Mycobact Dis. 1997 Jun;65(2):230-7. PMID 9251596
- [Background] Li HY, Hu LF, Huang WB, Liu GC, Yuan LC, Jin Z, Li X, Li JL, Yang ZM. Risk of relapse in leprosy after fixed-duration multidrug therapy. Int J Lepr Other Mycobact Dis. 1997 Jun;65(2):238-45. PMID 9251597
- [Background] Lockwood DN, Suneetha S. Leprosy: too complex a disease for a simple elimination paradigm. Bull World Health Organ. 2005 Mar;83(3):230-5. Epub 2005 Mar 16. PMID 15798849
- [Derived] Penna GO, Pontes MAA, Talhari S, Goncalves HS, Talhari C, Pessoa AS, Pedroza V, Buhrer-Sekula S, Stefani MMA, Penna MLF. Late relapses in leprosy patients in Brazil: 10-year post-trial of uniform multidrug therapy (U-MDT/CT-BR). Braz J Infect Dis. 2024 Mar-Apr;28(2):103745. doi: 10.1016/j.bjid.2024.103745. Epub 2024 Apr 30. PMID 38697216
- [Derived] Hungria EM, Buhrer-Sekula S, Oliveira RM, Aderaldo LC, Pontes MAA, Cruz R, de Goncalves HS, Penna MLF, Penna GO, Stefani MMA. Mycobacterium leprae-Specific Antibodies in Multibacillary Leprosy Patients Decrease During and After Treatment With Either the Regular 12 Doses Multidrug Therapy (MDT) or the Uniform 6 Doses MDT. Front Immunol. 2018 May 14;9:915. doi: 10.3389/fimmu.2018.00915. eCollection 2018. PMID 29867930
- [Derived] Penna GO, Buhrer-Sekula S, Kerr LRS, Stefani MMA, Rodrigues LC, de Araujo MG, Ramos AMC, de Andrade ARC, Costa MB, Rosa PS, Goncalves HS, Cruz R, Barreto ML, Pontes MAA, Penna MLF. Uniform multidrug therapy for leprosy patients in Brazil (U-MDT/CT-BR): Results of an open label, randomized and controlled clinical trial, among multibacillary patients. PLoS Negl Trop Dis. 2017 Jul 13;11(7):e0005725. doi: 10.1371/journal.pntd.0005725. eCollection 2017 Jul. PMID 28704363
- [Derived] Hungria EM, Buhrer-Sekula S, de Oliveira RM, Aderaldo LC, Pontes AA, Cruz R, Goncalves HS, Penna ML, Penna GO, Stefani MM. Leprosy reactions: The predictive value of Mycobacterium leprae-specific serology evaluated in a Brazilian cohort of leprosy patients (U-MDT/CT-BR). PLoS Negl Trop Dis. 2017 Feb 21;11(2):e0005396. doi: 10.1371/journal.pntd.0005396. eCollection 2017 Feb. PMID 28222139